CLINICAL TRIAL: NCT00971321
Title: Safety and Immunogenicity Study of GSK Biologicals' Pandemic Influenza Candidate Vaccine (GSK2340272A) in Children Aged 6 to 35 Months
Brief Title: Safety, Immunogenicity Study of GSK Biologicals' Pandemic Influenza Candidate Vaccine (H1N1) (GSK2340272A)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113462
Record Dates: First submitted 2009-08-27; First posted 2009-09-03 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2018-08

CONDITIONS: Influenza
Keywords: influenza infection; GSK Bio's influenza vaccine GSK2340272A
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- GSK 2340272A F1 Group (Experimental): Healthy male or female children, between and including 6 and 35 months of age, who received 2 doses of GSK2340272A Formulation 1 (F1) vaccine according to a 0, 21-day schedule, intramuscularly administered in the deltoid region of the arm or in the anterolateral region of the thigh if the subject was less than (<) 12 months at study entry.
  Interventions: Biological: Pandemic influenza vaccine GSK2340272A
- GSK 2340272A F2 Group (Experimental): Healthy male or female children, between and including 6 and 35 months of age, who received 2 doses of GSK2340272A Formulation 2 (F2) vaccine according to a 0, 21-day schedule, intramuscularly administered in the deltoid region of the arm or in the anterolateral region of the thigh if the subject was less than (<) 12 months at study entry.
  Interventions: Biological: Pandemic influenza vaccine GSK2340272A

INTERVENTIONS:
Biological: Pandemic influenza vaccine GSK2340272A — Two primary intramuscular (IM) injections

SUMMARY:
This trial is designed to assess the safety and immunogenicity of a prime-boost schedule of GSK Biologicals' investigational vaccine GSK2340272A in children aged between 6 and 35 months.

This protocol posting has been updated following protocol amendment 4, March 2010. The protocol posting sections impacted are number of subjects, primary and secondary endpoints and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol
* Children, male or female, aged between 6 and 35 months at the time of first study vaccination.
* Written informed consent obtained from the parent(s) or LAR(s) of the subject.
* Healthy children, as established by medical history and clinical examination when entering the study.
* Parent/LAR with access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user device.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period.
* Clinically or virologically confirmed influenza infection within six months preceding the study start.
* Planned administration of any vaccine 30 days prior and 30 days after any study vaccine administration.
* Chronic administration of immunosuppressants or other immune-modifying drugs within three months prior to enrolment in this study or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Acute or chronic, clinically-significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history and physical examination.
* History of hypersensitivity to vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment
* Administration of immunoglobulins and/or any blood products within the three months prior to the enrolment in this study, or planned during the study.
* Any condition which, in the opinion of the investigator, renders the subject unfit for participation in the study.
* Child in Care.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2009-09-10; Primary Completion 2010-11-24 (Actual); Study Completion 2010-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Spain (5):
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Garcia-Sicilia J, Aristegui J, Omenaca F, Carmona A, Tejedor JC, Merino JM, Garcia-Corbeira P, Walravens K, Bambure V, Moris P, Caplanusi A, Gillard P, Dieussaert I. Safety and persistence of the humoral and cellular immune responses induced by 2 doses of an AS03-adjuvanted A(H1N1)pdm09 pandemic influenza vaccine administered to infants, children and adolescents: Two open, uncontrolled studies. Hum Vaccin Immunother. 2015;11(10):2359-69. doi: 10.1080/21645515.2015.1063754. PMID 26176592
- [Derived] Carmona A, Omenaca F, Tejedor JC, Merino JM, Vaman T, Dieussaert I, Gillard P, Aristegui J. Immunogenicity and safety of AS03-adjuvanted 2009 influenza A H1N1 vaccine in children 6-35 months. Vaccine. 2010 Aug 16;28(36):5837-44. doi: 10.1016/j.vaccine.2010.06.065. Epub 2010 Jun 29. PMID 20600478
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 113462 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113462 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113462 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113462 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113462 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113462 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113462 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- GSK2340272A F1 Group: Healthy male or female children, between and including 6 and 35 months of age, who received 2 doses of GSK2340272A Formulation 1 (F1) vaccine according to a 0, 21-day schedule, intramuscularly administered in the deltoid region of the arm or in the anterolateral region of the thigh if the subject was less than (<) 12 months at study entry.
- GSK2340272A F2 Group: Healthy male or female children, between and including 6 and 35 months of age, who received 2 doses of GSK2340272A Formulation 2 (F2) vaccine according to a 0, 21-day schedule, intramuscularly administered in the deltoid region of the arm or in the anterolateral region of the thigh if the subject was less than (<) 12 months at study entry.
Period: Up to Day 42
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Started | 104 | 53
Completed | 104 | 53
Not Completed | 0 | 0
Period: Up to Month 7
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Started | 104 | 53
Completed | 100 | 51
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Migrated/moved from study area | 3 | 2
Period: Up to Month 11-12
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Started | 104 | 53
Completed | 99 | 50
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Migrated/moved from study area | 2 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group | Total
Number analyzed (Participants) | 104 | 53 | 157
Age, Continuous [Mean (Standard Deviation); unit: Months] | 19.3 (9.3) | 19.7 (8.8) | 19.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 26 | 69
  Male | 61 | 27 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage / African American | 1 | 0 | 1
  Geographic ancestry: American Indian or Alaskan Native | 1 | 0 | 1
  Geographic ancestry: White - Caucasian / European Heritage | 96 | 46 | 142
  Geographic ancestry: Other | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Seropositive Subjects for H1N1 Haemagglutination Inhibition (HI) Antibodies
Description: Seropositivity was defined as H1N1 HI antibody titers greater than or equal to (≥) 1:10. The strain assessed was Flu A/California/7/2009 (H1N1).
Time Frame: At Day 0
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 42, which included all evaluable subjects for whom assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after the second dose for all subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 101 | 48
Participants | 5 | 6

2. Primary Outcome: Number of Seropositive Subjects for H1N1 Haemagglutination Inhibition (HI) Antibodies
Description: as for outcome 1
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 97 | 50
Participants | 97 | 50

3. Primary Outcome: Titers for H1N1 Haemagglutination Inhibition (HI) Antibodies
Description: Antibody titers are presented as geometric mean titers (GMTs), with a reference seropositivity cut-off value greater than or equal to (≥) 1:10. The strain assessed was Flu A/California/7/2009 (H1N1).
Time Frame: At Day 0
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 42, which included all evaluable subjeects for whom assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after the second dose for all subjects.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 101 | 48
Titers | 5.75 [5.00 to 6.63] | 6.82 [5.22 to 8.91]

4. Primary Outcome: Titers for H1N1 Haemagglutination Inhibition (HI) Antibodies
Description: as for outcome 3
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 97 | 50
Titers | 2007.70 [1805.24 to 2232.87] | 2259.61 [1947.61 to 2621.59]

5. Primary Outcome: Number of Seroconverted Subjects in Terms of H1N1 Haemagglutination Inhibition (HI) Antibodies
Description: Seroconversion (SCR) was defined as the percentage of vaccinees that have either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The strain assessed was Flu A/California/7/2009 (H1N1).
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 97 | 48
Participants | 97 | 48

6. Primary Outcome: Number of Seroprotected Subjects for H1N1 Haemagglutination Inhibition (HI) Antibodies
Description: Seroprotection (SPR) was defined as the percentage of vaccinees with a serum HI titer ≥ 1:40 that usually is accepted as indicating protection. The strain assessed was Flu A/California/7/2009 (H1N1).
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 97 | 50
Participants | 97 | 50

7. Primary Outcome: Seroconversion Factor (SCF) for H1N1 Haemagglutination Inhibition (HI) Antibody Titers
Description: Seroconversion factor was defined as the fold increase in serum HI geometric mean titers (GMTs) post-vaccination compared to pre-vaccination. The strain assessed was Flu A/California/7/2009 (H1N1).
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 97 | 48
Fold change | 346.86 [287.54 to 418.42] | 322.67 [231.61 to 449.52]

8. Secondary Outcome: Number of Seropositive Subjects for H1N1 Haemagglutination Inhibition (HI) Antibodies
Description: as for outcome 1
Time Frame: At Days 0, 21, 42, and at Month 11-12
Population: The ATP cohort for antibody persistence at Month 11-12 included all evaluable subjects who had received at least one dose of vaccine according to their treatment assignment and for whom data concerning immunogenicity outcome measures and assay results were available for antibodies against the study vaccine component at Month 11-12.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 83 | 37
Participants
  Flu A/CAL/7/2009, Day 0 | 4 | 4
  Flu A/CAL/7/2009, Day 21 | 83 | 37
  Flu A/CAL/7/2009, Day 42 | 83 | 37
  Flu A/CAL/7/2009, Month 11-12 | 83 | 37

9. Secondary Outcome: Titers for H1N1 Haemagglutination Inhibition (HI) Antibodies
Description: as for outcome 3
Time Frame: At Days 0, 21, 42 and at Month 11-12
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 83 | 37
Titers
  Flu A/CAL/7/2009, Day 0 | 5.8 [5.0 to 6.8] | 6.2 [5.0 to 7.8]
  Flu A/CAL/7/2009, Day 21 | 234.0 [202.9 to 269.8] | 255.5 [205.4 to 317.9]
  Flu A/CAL/7/2009, Day 42 | 1758.0 [1553.8 to 1989.1] | 1879.2 [1504.2 to 2347.7]
  Flu A/CAL/7/2009, Month 11-12 | 212.5 [182.8 to 247.0] | 239.3 [201.6 to 284.0]

10. Secondary Outcome: Number of Seroconverted Subjects in Terms of H1N1 Haemagglutination Inhibition (HI) Antibody Titers
Description: as for outcome 5
Time Frame: At Days 21, 42 and at Month 11-12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 83 | 37
Participants
  Flu A/CAL/7/2009, Day 21 | 82 | 37
  Flu A/CAL/7/2009, Day 42 | 83 | 37
  Flu A/CAL/7/2009, Month 11-12 | 81 | 36

11. Secondary Outcome: Number of Seroprotected Subjects for H1N1 Haemagglutination Inhibition (HI) Antibodies
Description: as for outcome 6
Time Frame: At Days 0, 21, 42 and at Month 11-12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 83 | 37
Participants
  Flu A/CAL/7/2009, Day 0 | 3 | 3
  Flu A/CAL/7/2009, Day 21 | 83 | 37
  Flu A/CAL/7/2009, Day 42 | 83 | 37
  Flu A/CAL/7/2009, Month 11-12 | 83 | 37

12. Secondary Outcome: Seroconversion Factor (SCF) for H1N1 Haemagglutination Inhibition (HI) Antibody Titers
Description: as for outcome 7
Time Frame: At Days 21, 42 and at Month 11-12
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 83 | 37
Fold change
  Flu A/CAL/7/2009, Day 21 | 40.3 [34.3 to 47.2] | 41.2 [32.2 to 52.7]
  Flu A/CAL/7/2009, Day 42 | 302.5 [248.2 to 368.7] | 302.8 [211.8 to 432.9]
  Flu A/CAL/7/2009, Month 11-12 | 36.6 [30.0 to 44.6] | 38.6 [29.5 to 50.4]

13. Secondary Outcome: Titers for Serum Neutralising Antibodies
Description: Antibody titers are presented as geometric mean titers (GMTs), with a reference seropositivity cut-off value greater than or equal to (≥) 1:8. The strain assessed was Flu A/Neth/602/09.
Time Frame: At Days 0, 21 and 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after the second dose for all subjects.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 65 | 32
Titers
  Flu A/Neth/602/2009, Day 0: number analyzed (Participants) | 65 | 30
  Flu A/Neth/602/2009, Day 0 | 5.35 [3.94 to 7.26] | 5.40 [3.76 to 7.77]
  Flu A/Neth/602/2009, Day 21: number analyzed (Participants) | 62 | 30
  Flu A/Neth/602/2009, Day 21 | 37.88 [26.46 to 54.22] | 51.23 [29.85 to 87.90]
  Flu A/Neth/602/2009, Day 42: number analyzed (Participants) | 63 | 32
  Flu A/Neth/602/2009, Day 42 | 1488.85 [1144.23 to 1937.25] | 1907.39 [1250.94 to 2908.34]

14. Secondary Outcome: Titers for Serum Neutralising Antibodies
Description: as for outcome 13
Time Frame: At Days 0, 21, 42 and at Month 11-12
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 57 | 24
Titers
  Flu A/Neth/602/09, Day 0 | 5.6 [3.9 to 7.9] | 5.7 [3.6 to 8.9]
  Flu A/Neth/602/09, Day 21: number analyzed (Participants) | 53 | 23
  Flu A/Neth/602/09, Day 21 | 36.9 [24.5 to 55.4] | 50.8 [25.6 to 100.7]
  Flu A/Neth/602/09, Day 42: number analyzed (Participants) | 54 | 23
  Flu A/Neth/602/09, Day 42 | 1416.1 [1048.1 to 1913.3] | 1960.6 [1097.0 to 3504.0]
  Flu A/Neth/602/09, Month 11-12: number analyzed (Participants) | 49 | 22
  Flu A/Neth/602/09, Month 11-12 | 312.8 [223.1 to 438.6] | 444.4 [286.5 to 689.3]

15. Secondary Outcome: Number of Subjects With Vaccine Response for Serum Neutralising Antibodies
Description: Vaccine response rate was defined as the percentage of vaccinees with a minimum 4-fold increase in titer at post-vaccination for neutralising antibody response. For initially seronegative subjects, antibody titer ≥ 1:32 after vaccination; For initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The strain assessed was Flu A/Neth/602/2009.
Time Frame: At Days 21 and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 61 | 29
Participants
  Flu A/Neth/602/2009, Day 21: number analyzed (Participants) | 59 | 29
  Flu A/Neth/602/2009, Day 21 | 34 | 18
  Flu A/Neth/602/2009, Day 42 | 60 | 29

16. Secondary Outcome: Number of Subjects With Vaccine Response for Serum Neutralising Antibodies
Description: as for outcome 15
Time Frame: At Days 21, 42 and at Month 11-12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 25 | 12
Participants
  Flu A/Neth/602/2009, Day 21 | 14 | 8
  Flu A/Neth/602/2009, Day 42 | 24 | 12
  Flu A/Neth/602/2009, Month 11-12: number analyzed (Participants) | 22 | 10
  Flu A/Neth/602/2009, Month 11-12 | 19 | 10

17. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period after each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 104 | 53
Participants
  Any Pain, Dose 1 | 37 | 31
  Grade 3 Pain, Dose 1 | 1 | 0
  Any Redness, Dose 1 | 19 | 17
  Grade 3 Redness, Dose 1 | 0 | 2
  Any Swelling, Dose 1 | 12 | 11
  Grade 3 Swelling, Dose 1 | 0 | 1
  Any Pain, Dose 2: number analyzed (Participants) | 104 | 52
  Any Pain, Dose 2 | 43 | 27
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 104 | 52
  Grade 3 Pain, Dose 2 | 3 | 2
  Any Redness, Dose 2: number analyzed (Participants) | 104 | 52
  Any Redness, Dose 2 | 34 | 23
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 104 | 52
  Grade 3 Redness, Dose 2 | 1 | 6
  Any Swelling, Dose 2: number analyzed (Participants) | 104 | 52
  Any Swelling, Dose 2 | 30 | 17
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 104 | 52
  Grade 3 Swelling, Dose 2 | 1 | 4
  Any Pain, Across doses | 54 | 37
  Grade 3 Pain, Across doses | 4 | 2
  Any Redness, Across doses | 41 | 27
  Grade 3 Redness, Across doses | 1 | 6
  Any Swelling, Across doses | 38 | 21
  Grade 3 Swelling, Across doses | 1 | 5

18. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 loss of appetite= not eating at all. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period after each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who has their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 104 | 53
Participants
  Any Drowsiness, Dose 1 | 24 | 14
  Grade 3 Drowsiness, Dose 1 | 0 | 2
  Related Drowsiness, Dose 1 | 17 | 11
  Any Irritability, Dose 1 | 33 | 17
  Grade 3 Irritability, Dose 1 | 2 | 5
  Related Irritability, Dose 1 | 28 | 12
  Any Loss of appetite, Dose 1 | 25 | 17
  Grade 3 Loss of appetite, Dose 1 | 1 | 1
  Related Loss of appetite, Dose 1 | 18 | 11
  Any Fever, Dose 1 | 21 | 13
  Grade 3 Fever, Dose 1 | 1 | 1
  Related Fever, Dose 1 | 16 | 10
  Any Drowsiness, Dose 2: number analyzed (Participants) | 104 | 52
  Any Drowsiness, Dose 2 | 36 | 25
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 104 | 52
  Grade 3 Drowsiness, Dose 2 | 0 | 2
  Related Drowsiness, Dose 2: number analyzed (Participants) | 104 | 52
  Related Drowsiness, Dose 2 | 35 | 22
  Any Irritability, Dose 2: number analyzed (Participants) | 104 | 52
  Any Irritability, Dose 2 | 48 | 31
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 104 | 52
  Grade 3 Irritability, Dose 2 | 3 | 4
  Related Irritability, Dose 2: number analyzed (Participants) | 104 | 52
  Related Irritability, Dose 2 | 45 | 27
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 104 | 52
  Any Loss of appetite, Dose 2 | 44 | 30
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 104 | 52
  Grade 3 Loss of appetite, Dose 2 | 4 | 4
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 104 | 52
  Related Loss of appetite, Dose 2 | 41 | 26
  Any Fever, Dose 2: number analyzed (Participants) | 104 | 52
  Any Fever, Dose 2 | 70 | 37
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 104 | 52
  Grade 3 Fever, Dose 2 | 4 | 9
  Related Fever, Dose 2: number analyzed (Participants) | 104 | 52
  Related Fever, Dose 2 | 64 | 34
  Any Drowsiness, Across doses | 47 | 31
  Grade 3 Drowsiness, Across doses | 0 | 3
  Related Drowsiness, Across doses | 43 | 26
  Any Irritability, Across doses | 60 | 38
  Grade 3 Irritability, Across doses | 5 | 8
  Related Irritability, Across doses | 54 | 31
  Any Loss of appetite, Across doses | 54 | 35
  Grade 3 Loss of appetite, Across doses | 5 | 5
  Related Loss of appetite, Across doses | 49 | 29
  Any Fever, Across doses | 79 | 41
  Grade 3 Fever, Across doses | 5 | 10
  Related Fever, Across doses | 70 | 37

19. Secondary Outcome: Number of Subjects With Any Medically-attended Events (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.
Time Frame: During the entire study period (Day 0 up to Month 7 and Day 0 up to Month 11-12)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 104 | 53
Participants
  Any MAEs, up to Month 7 | 92 | 40
  Any MAEs, up to Month 11-12 | 94 | 45

20. Secondary Outcome: Number of Subjects With Any Adverse Events of Specific Interest (AESIs)/ Potential Immune-mediated Disease (pIMDs)
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration. Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: During the entire study period (Day 0 up to Month 11-12)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 104 | 53
Participants | 0 | 0

21. Secondary Outcome: Number of Subjects With Normal/Abnormal Biochemical Levels
Description: Among biochemical parameters assessed were: alanine aminotrasferase [ALAT], aspartate aminotransferase [ASAT], bilirubin total [BIL/T], bilirubin direct [BIL/D], creatinine [CREA] and blood urea nitrogen [BUN]. Levels of biochemical parameters assessed with respect to normal laboratory values were - unknown, below, within and above.
Time Frame: At Days 0, 21 and 42
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 104 | 53
Participants
  ALAT, Day 0: Unknown | 3 | 4
  ALAT, Day 0: Below | 0 | 0
  ALAT, Day 0: Within | 101 | 49
  ALAT, Day 0: Above | 0 | 0
  ALAT, Day 21: number analyzed (Participants) | 104 | 52
  ALAT, Day 21: Unknown | 1 | 1
  ALAT, Day 21: Below | 0 | 0
  ALAT, Day 21: Within | 100 | 50
  ALAT, Day 21: Above | 3 | 1
  ALAT, Day 42: number analyzed (Participants) | 103 | 53
  ALAT, Day 42: Unknown | 1 | 0
  ALAT, Day 42: Below | 0 | 0
  ALAT, Day 42: Within | 98 | 53
  ALAT, Day 42: Above | 4 | 0
  ASAT, Day 0: Unknown | 3 | 3
  ASAT, Day 0: Below | 0 | 0
  ASAT, Day 0: Within | 100 | 49
  ASAT, Day 0: Above | 1 | 1
  ASAT, Day 21: number analyzed (Participants) | 104 | 52
  ASAT, Day 21: Unknown | 4 | 3
  ASAT, Day 21: Below | 0 | 0
  ASAT, Day 21: Within | 94 | 48
  ASAT, Day 21: Above | 6 | 1
  ASAT, Day 42: number analyzed (Participants) | 103 | 53
  ASAT, Day 42: Unknown | 1 | 0
  ASAT, Day 42: Below | 0 | 0
  ASAT, Day 42: Within | 96 | 53
  ASAT, Day 42: Above | 6 | 0
  BIL/T, Day 0: Unknown | 3 | 4
  BIL/T, Day 0: Below | 0 | 0
  BIL/T, Day 0: Within | 101 | 49
  BIL/T, Day 0: Above | 0 | 0
  BIL/T, Day 21: number analyzed (Participants) | 104 | 52
  BIL/T, Day 21: Unknown | 2 | 1
  BIL/T, Day 21: Below | 0 | 0
  BIL/T, Day 21: Within | 102 | 51
  BIL/T, Day 21: Above | 0 | 0
  BIL/T, Day 42: number analyzed (Participants) | 103 | 53
  BIL/T, Day 42: Unknown | 1 | 0
  BIL/T, Day 42: Below | 0 | 0
  BIL/T, Day 42: Within | 102 | 53
  BIL/T, Day 42: Above | 0 | 0
  BIL/D, Day 0: Unknown | 3 | 4
  BIL/D, Day 0: Below | 0 | 0
  BIL/D, Day 0: Within | 101 | 49
  BIL/D, Day 0: Above | 0 | 0
  BIL/D, Day 21: number analyzed (Participants) | 104 | 52
  BIL/D, Day 21: Unknown | 1 | 1
  BIL/D, Day 21: Below | 0 | 0
  BIL/D, Day 21: Within | 103 | 51
  BIL/D, Day 21: Above | 0 | 0
  BIL/D, Day 42: number analyzed (Participants) | 103 | 53
  BIL/D, Day 42: Unknown | 1 | 0
  BIL/D, Day 42: Below | 0 | 0
  BIL/D, Day 42: Within | 102 | 53
  BIL/D, Day 42: Above | 0 | 0
  CREA, Day 0: Unknown | 3 | 3
  CREA, Day 0: Below | 32 | 16
  CREA, Day 0: Within | 67 | 34
  CREA, Day 0: Above | 2 | 0
  CREA, Day 21: number analyzed (Participants) | 104 | 52
  CREA, Day 21: Unknown | 1 | 2
  CREA, Day 21: Below | 34 | 19
  CREA, Day 21: Within | 69 | 30
  CREA, Day 21: Above | 0 | 1
  CREA, Day 42: number analyzed (Participants) | 103 | 53
  CREA, Day 42: Unknown | 1 | 0
  CREA, Day 42: Below | 37 | 16
  CREA, Day 42: Within | 65 | 37
  CREA, Day 42: Above | 0 | 0
  BUN, Day 0: Unknown | 3 | 4
  BUN, Day 0: Below | 1 | 0
  BUN, Day 0: Within | 77 | 36
  BUN, Day 0: Above | 23 | 13
  BUN, Day 21: number analyzed (Participants) | 104 | 52
  BUN, Day 21: Unknown | 1 | 1
  BUN, Day 21: Below | 0 | 0
  BUN, Day 21: Within | 79 | 37
  BUN, Day 21: Above | 24 | 14
  BUN, Day 42: number analyzed (Participants) | 103 | 53
  BUN, Day 42: Unknown | 1 | 0
  BUN, Day 42: Below | 1 | 0
  BUN, Day 42: Within | 76 | 41
  BUN, Day 42: Above | 25 | 12

22. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During a 21 day follow-up period after the first vaccination and during a 62-day follow-up period after the second vaccination (Days 0 - 84)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 104 | 53
Participants
  Any AE(s) | 98 | 47
  Grade 3 AE(s) | 18 | 8
  Related AE(s) | 12 | 8

23. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (Day 0 up to Month 11-12)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group
Number analyzed (Participants) | 104 | 53
Participants | 2 | 6

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: during a 21 day follow-up period after the first vaccination and during a 62-day follow-up period after the second vaccination (Days 0 - 84); SAEs: during the entire study period (Day 0 up to Month 11-12).
Arm/Group | GSK 2340272A F1 Group | GSK 2340272A F2 Group
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/53
Serious Adverse Events (participants affected / at risk) | 2/104 | 6/53
Other Adverse Events (participants affected / at risk) | 103/104 | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK 2340272A F1 Group (N=104) | GSK 2340272A F2 Group (N=53)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK 2340272A F1 Group (N=104) | GSK 2340272A F2 Group (N=53)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6)
Bronchitis (Infections and infestations) | 12 (14) | 6 (7)
Conjunctivitis (Infections and infestations) | 6 (6) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 7 (8)
Decreased appetite (Metabolism and nutrition disorders) | 54 (69) | 35 (47)
Diarrhoea (Gastrointestinal disorders) | 15 (16) | 7 (8)
Erythema (Skin and subcutaneous tissue disorders) | 41 (53) | 27 (40)
Gastroenteritis (Infections and infestations) | 12 (14) | 8 (11)
Irritability (Psychiatric disorders) | 61 (83) | 38 (48)
Laryngitis (Infections and infestations) | 6 (7) | 3 (3)
Otitis media (Infections and infestations) | 6 (7) | 3 (3)
Otitis media acute (Infections and infestations) | 9 (10) | 1 (2)
Pain (General disorders) | 54 (80) | 37 (58)
Pharyngitis (Infections and infestations) | 11 (13) | 2 (2)
Pyrexia (General disorders) | 81 (100) | 43 (55)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0)
Respiratory tract infection (Infections and infestations) | 5 (6) | 3 (3)
Rhinitis (Infections and infestations) | 4 (4) | 3 (4)
Somnolence (Nervous system disorders) | 47 (60) | 31 (39)
Swelling (General disorders) | 38 (42) | 21 (28)
Tonsillitis (Infections and infestations) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 59 (90) | 24 (34)
Vomiting (Gastrointestinal disorders) | 6 (7) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.